CLINICAL TRIAL: NCT05167903
Title: The Effect of Time-restricted Eating Combined With Exercise Training on Body Composition and Cardiometabolic Health; Randomized Controlled Trial (TERA)
Brief Title: The Effect of Time-restricted Eating Combined With Exercise Training on Body Composition and Cardiometabolic Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Gepner Yftach, Principal Investigator, Tel Aviv University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0057-21-ASF
Record Dates: First submitted 2021-10-26; First posted 2021-12-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Metabolic Syndrome
Keywords: Time-restricted eating; muscle mass; strength; cardio-metabolic risk
MeSH Terms: conditions — Metabolic Syndrome; Intermittent Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time-restricted eating (Experimental): Participants in the TRE group will be instructed to consume all meals between 12pm to 8pm (8 h eating window with 16 h of fasting)
  Interventions: Behavioral: Time-restricted eating
- Normal Diet (ND) (Experimental): The ND group will consume all meals between 6 am - 10 pm (16 h eating window with 8 h of fasting, ad-libitum)
  Interventions: Other: Normal Diet

INTERVENTIONS:
Other: Normal Diet — All praticipants in ND will perform supervised and monitored RT three time per week for the 10 weeks of intervention. The ND group will consume all meals between 6 am - 10 pm (16 h eating window with 8 h of fasting, ad-libitum).
  Other Names: ND
  Arms: Normal Diet (ND)
Behavioral: Time-restricted eating — All participants in TRE will perform supervised and monitored RT three time per week for the 10 weeks of intervention. Participants in the TRE group will be instructed to consume all meals between 12pm to 8pm, and to avoid consumption of food or caloric drinks during the fasting period (8 h eating window with 16 h of fasting).
  Other Names: TRE
  Arms: Time-restricted eating

SUMMARY:
The aim of the study is to determine the effect of resistance training (RT) combined with time-restricted eating (TRE) or normal diet (ND) on muscle mass, and strength. Additionally, the study will compare between TRE and ND and its effects on cardiometabolic health, mitochondria function and body composition among people with metabolic syndrome.

In this randomized controlled trial, 50 males with metabolic syndrome (elevated waist circumference, blood pressure, triglycerides, fasting glucose and low high-density lipoprotein cholesterol) between the age of 40-60y and with BMI between 25-33 kg/m2 will be randomized to either TRE+RT (n=25) or ND+RT (n=25). All participants will perform supervised and monitored RT three time per week for the 10 weeks of intervention Study measurements; Changes in body composition, muscle mass and adipose tissue distribution will be measured by 3-Tesla magnetic resonance imaging (MRI), dual energy x-ray absorptiometry (DXA), air displacement plethysmography (BODPOD) and Bioelectrical Impedance analysis (BIA). Muscular Strength will be assessed. Blood samples, including lipid and glycemic profile. muscle biopsy taken from the vastus lateralis muscle.

DETAILED DESCRIPTION:
Primary aim. Determine the effect of TRE or ND, combined with RT training, on muscle mass and strength as adaptive response to 10 weeks of intervention among people with metabolic syndrome.

Secondary aims. Determine the effect of TRE combined with RT on cardiometabolic health lipid profile and HbA1C (C), Mitochondria function and oxygen consumption (D) and Body composition assessment (E).

ELIGIBILITY:
Inclusion Criteria:

* Subject with metabolic syndrome
* BMI between 25-33 kg/m²
* Age 40-60
* Without cardiac and pulmonary disease
* Did not engage exercise training in the last year.
* Willing and able to read, understand and sign an informed consent

Exclusion Criteria:

* Participants that have cardiopulmonary disease
* Inability to attend scheduled clinic visits and/or comply with the study protocol
* Active smokers
* Previous regular exercise training in the previous yea
* Major orthopedic injury at the past 3 months
* Inability to perform an MRI (due to claustrophobia, or metal in their body)
* Subjects that uses drugs that affect muscle metabolism

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Self-representation of gender identity.
Enrollment: 50 (Estimated)
Dates: Start 2022-05-15 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Primary aim muscle mass | 10 weeks
  Muscle mass volume using MRI (cm3)
Primary aim free fat mass | 10 weeks
  Free fat mass will be mesured in in kg using DXA , BOD POD and BIA
Primary aim Maximum strength | 10 weeks
  Maximum strength by one-repetition maximum (kg) using two exercise (bench press, hack squat)

SECONDARY OUTCOMES:
Secondary aims Cardiometabolic profile | 10 weeks
  Cardiometabolic profile [glucose (mg/dl), total cholesterol (mg/dl), HDL (mg/dl), LDL (mg/dl), TG (mg/dl)] will be mesured using blood test
Secondary aims body composition assessment | 10 weeks
  Body composition assessment fat mass (kg) using DXA, BOD POD and BIA

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv University, Tel Aviv, Other, Israel

IPD SHARING:
Plan to Share IPD: No